CLINICAL TRIAL: NCT01740843
Title: The Effect of tDCS on Motor Performance and Cortical Excitability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Koen Cuypers, Drs. Koen Cuypers, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MECU2012-004
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Cortical Excitability; Motor Performance; tDCS
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low intensity anodal tDCS (Active Comparator): tDCS will be administered for 10 min at 1mA
  Interventions: Device: transcranial direct current stimulation (tDCS) (NeuroConn DC-stimulator)
- High intensity anodal tDCS (Experimental): tDCS will be administered for 10 min at 2.5mA
  Interventions: Device: transcranial direct current stimulation (tDCS) (NeuroConn DC-stimulator)
- Sham tDCS (Sham Comparator): Sham will be administered for 10 min at 0 mA
  Interventions: Device: transcranial direct current stimulation (tDCS) (NeuroConn DC-stimulator)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) (NeuroConn DC-stimulator) — The anode is fixed on the primary cortex and the cathode will be fixed on the contralateral supraorbital region.
  Other Names: NeuroConn DC-stimulator

SUMMARY:
In this study the effect of tDCS intensity on motor performance and corticospinal (CS) excitability is evaluated. The investigators expect that a positive relationship between current intensity and motor performance/CS excitability.

ELIGIBILITY:
Inclusion Criteria:

- Healthy subjects

Exclusion Criteria:

* Contraindications for tDCS/TMS
* TMS measurements have to be possible

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in motor performance | Baseline and POST (30 min after baseline) intervention
  motor performance is assessed using different reaction time paradigms (simple reaction time, choice reaction time). This is done at baseline and immediately after the intervention (30 min after baseline)
Change in cortical excitability | Baseline and POST (30 min after baseline) intervention
  Cortical excitability is measured using trancranial magnetic stimulation (TMS) measuring muscle evoked potentials (MEPs) at baseline and POST (30 min after baseline).